CLINICAL TRIAL: NCT04057846
Title: EUS-guided Drainage of Large Walled-off Pancreatic Necrosis Using Lumen Apposing Metal Stents or Standard Double Pigtail Technique. A Single-center, Open-label, Randomized, Superiority Trial
Brief Title: Lumen Apposing Metal Stents vs Double Pigtail Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Gasdal Karstensen (Other)
Responsible Party: Sponsor-Investigator, John Gasdal Karstensen, Principal Investigator, MD, PhD, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAMS vs DPT
Record Dates: First submitted 2019-07-29; First posted 2019-08-15 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Pancreatitis,Acute Necrotizing
Keywords: Walled of necrosis; Endoscopic drainage; Lumen apposing metal stents
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Intervention Model Description: A single-center, open-label, randomized, superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Double pigtail (Active Comparator): Plastic stent group EUS-guided drainage shall be performed as follows: a) Puncture of WON with a 19 GA Access needle (Cook Medical), b) aspiration of fluid in WON for microbiological assessment, c) insertion of guidewire (0.035 inch, 450 cm, Dreamwire (Boston Scientific), d) creation of transmural tract with needle knife over the guidewire, e) dilatation of tract to a diameter of 15 mm with dilation balloon (EZDilate, Olympus), f) insertion of two 7-Fr/6 cm double pigtail stents and a 7-Fr naso-cystic irrigation catheter.
  Interventions: Device: EUS guided transgastric drainage
- Lumen apposing metal stent (Experimental): LAMS shall be the Hot AXIOS stent with electrocautery-enhanced delivery system (Boston Scientific). The stent is a through-the-scope, fully covered, self-expandable metal stents with a diameter of 20 mm and a length of 10 mm. Before placement of the LAMS, the WON shall be punctured with a 19 GA Access needle (Cook Medical) and fluid in WON aspirated for microbiological assessment. Thereafter the LAMS shall be placed as follows: After directly puncturing the WON using the electrocautery tip (without the use of a guidewire to assist in stent insertion), the delivery catheter is advanced into the WON and the distal flange is deployed under EUS-guidance. The proximal flange is then released under EUS guidance or endoscopic view. After placement of the LAMS, a 7-Fr/4cm double pigtail and a 7-Fr nasocystic irrigation catheter shall be placed through the LAMS.
  Interventions: Device: EUS guided transgastric drainage

INTERVENTIONS:
Device: EUS guided transgastric drainage — Whenever possible, randomisation and intervention shall be postponed until 4 weeks after onset of pancreatitis in line with international guidelines. All procedures in this study shall be performed by three experienced endoscopists (PNS, EFH, SN), who all have an extensive experience in endoscopic ultrasound (EUS-) guided drainage of pancreatic collections and the use of self-expanding stents. They have together performed more than 300 endoscopic, transmural drainage and debridement procedures in patients with WON since 2005. Endosonography-guided, transgastric drainage of the WONs shall be performed using a curve-linear echoendoscope (endoscope: Olympus GF-UCT180; ultrasound scanner: Hitachi Arietta 850 or Olympus EU-ME2). All collections shall be treated by single tract transmural cystogastrostomy (single-gate technique). T

SUMMARY:
While the majority of patients with acute pancreatitis suffer a mild and uncomplicated course of disease, up to 20% develop a more severe course with development of pancreatic and/or peripancreatic necroses. With time, these necroses become encapsulated with a well-defined inflammatory wall, so called walled-off necroses (WON). Up to 30% of WONs become infected, which prolongs the length of hospital stay, increases morbidity and mortality significantly, and generally requires an invasive intervention. During the last decade, minimally invasive therapies consisting of percutaneous and endoscopic, transluminal drainage followed, if necessary, by percutaneous or endoscopic necrosectomy, have replaced open surgery as the standard treatment resulting in better patient outcomes. The investigators have for nearly two decades been practicing an endoscopic step-up approach as standard treatment for infected WON.

Recently, lumen apposing metal stents (LAMS) have been introduced for the treatment of pancreatic fluid collections. The stent is fully-covered and shaped with two bilateral anchor flanges with a saddle in between. A dedicated through-the-scope delivery system, where the tip serves as an electro cautery device enables extra-luminal access and deployment of the stent. Initial results from primarily retrospective case series were promising. However, a recent randomized controlled trial failed to demonstrate superiority in terms of number of necrosectomies needed, treatment success, clinical adverse events, readmissions, length of hospital stay (LOS), and overall treatment costs. Furthermore, a number of serious adverse events with development of pseudoaneurisms probably due to collapse of the cavity have led to alterations in treatment with sequential computed tomography (CT) scans and insertion of double pigtail stents within the metal stent. In that trial, the mean diameter of the treated necroses was limited and in addition, the study was launched before the introduction of a novel 20 mm in diameter LAMS. The investigators hypothesize, that use of a 20 mm LAMS in large caliber WON is superior to the standard double pigtail technique.

Aim To compare the use of a novel 20 mm lumen apposing metal stent (LAMS) (Hot Axios, Boston Scientific) with a conventional double pigtail technique for endoscopic transluminal drainage of large (> 15 cm) pancreatic and/or peripancreatic walled-of necrosis (WON).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (all criteria must be fulfilled):

1. Patients with acute, necrotizing pancreatitis and

   1. WON exceeding a diameter of 15 cm (measured on contrast-enhanced CT (CECT); see details on imaging tests below). WON is defined based on the revised Atlanta criteria as a mature, encapsulated pancreatic or peripancreatic necrosis with a well-defined inflammatory wall[12].
   2. Imaging test(s) must be done within 1 week before the index drainage procedure.
   3. Debut of pancreatitis must be within 3 months before the index drainage procedure.
2. One or more indication(s) for endoscopic, transmural drainage must be established:

1. Confirmed or suspected infection.1 2. Severe intraabdominal hypertension or abdominal compartment syndrome. 3. Persisting abdominal pain, early satiety, or general discomfort. 4. Obstruction of the GI or biliary tract. 5. Leakage of pancreatic juice, e.g. ascites or pleural effusion.

3. Preoperatively, the WON must be considered eligible for endoscopic, transgastric drainage with both conventional double pigtail and LAMS technique. Distance between the gastric wall and WON must not exceed one cm and there must be no major interposed vessels.

Infection in WON:

1. Confirmed infected necrosis is defined as a) positive culture from WON obtained by fine- needle aspiration prior to or at the first drainage procedure or b) presence of gas in WON on CECT prior to drainage with no earlier puncture/drainage and no signs of perforation to the GI tract.
2. Infected necrosis is suspected when a patient with WON present with clinical signs of persistent sepsis without other causes of infection.

Exclusion Criteria:

1. Patients under the age of 18.
2. Pregnancy.
3. Known or suspected malignant disease.
4. Pancreatitis secondary to trauma or surgical intervention.
5. Chronic pancreatitis.
6. Collections that may only be drained from the duodenum.
7. Previous surgical or endoscopic drainage or necrosectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Number of necrosectomies | Through study completion, an average of 2 year
  Number of debridement procedures (endoscopic and video-assisted) needed throughout the disease course.

SECONDARY OUTCOMES:
Number of endoscopic procedures | Through study completion, an average of 6 months
  Number of endoscopic procedures (drainage (including redilatation) and debridement)
Total number of drainage and debridement procedures (radiological, endoscopic, and surgical) | Through study completion, an average of 6 months
Number of days from index drainage procedure until removal of naso-cystic catheter | Through study completion, an average of 6 months
Duration of drainage and debridement procedures | Through study completion, an average of 6 months
  Duration of drainage and debridement procedures (index and cumulated). It will be in minutes
Length of hospital stay from the index drainage procedure | Through study completion, an average of 6 months
  Days of hospital stay from the index drainage procedure
Length of ICU stay | Through study completion, an average of 6 months
  Days in the ICU
Resolution of pre-interventional systemic inflammatory response syndrome (SIRS) (sepsis) | Through study completion, an average of 6 months
  Restoration of normal blood pressure, temperature, heart rate, inspiratory rate, and white blod cell count
New onset episodes of culture verified bacteremia | Through study completion, an average of 6 months
Occurrence of splanchnic vein thrombosis (portal-, splenic-, or superior mesenteric vein) | Through study completion, an average of 6 months
Need for tube feeding (naso-gastric or naso-jejunal) or parenteral nutrition | Through study completion, an average of 6 months
CRP-area under curve (AUC) from the index drainage procedure until discharge from hospital | Though the hospital stay, an average of 6 months
Number of adverse events according to the ASGE lexicon and Clavien-Dindo. | Though the hospital stay, an average of 6 months
  Specific adverse events and grouped by severity
Mortality | Though the hospital stay, an average of 6 months
  The rate mortality compared between the two study groups
Exocrine and endocrine insufficiency | Though the hospital stay, an average of 6 months
  The unset of diabetes and Steatorré
Total treatment costs. | Through study completion
  In euros and dollars

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Capital, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Dijk SM, Hallensleben NDL, van Santvoort HC, Fockens P, van Goor H, Bruno MJ, Besselink MG; Dutch Pancreatitis Study Group. Acute pancreatitis: recent advances through randomised trials. Gut. 2017 Nov;66(11):2024-2032. doi: 10.1136/gutjnl-2016-313595. Epub 2017 Aug 24. PMID 28838972
- [Background] Banks PA, Freeman ML; Practice Parameters Committee of the American College of Gastroenterology. Practice guidelines in acute pancreatitis. Am J Gastroenterol. 2006 Oct;101(10):2379-400. doi: 10.1111/j.1572-0241.2006.00856.x. No abstract available. PMID 17032204
- [Background] Yan L, Dargan A, Nieto J, Shariaha RZ, Binmoeller KF, Adler DG, DeSimone M, Berzin T, Swahney M, Draganov PV, Yang DJ, Diehl DL, Wang L, Ghulab A, Butt N, Siddiqui AA. Direct endoscopic necrosectomy at the time of transmural stent placement results in earlier resolution of complex walled-off pancreatic necrosis: Results from a large multicenter United States trial. Endosc Ultrasound. 2019 May-Jun;8(3):172-179. doi: 10.4103/eus.eus_108_17. PMID 29882517
- [Background] Schmidt PN, Novovic S, Roug S, Feldager E. Endoscopic, transmural drainage and necrosectomy for walled-off pancreatic and peripancreatic necrosis is associated with low mortality--a single-center experience. Scand J Gastroenterol. 2015 May;50(5):611-8. doi: 10.3109/00365521.2014.946078. Epub 2015 Feb 3. PMID 25648776
- [Background] Bang JY, Navaneethan U, Hasan MK, Sutton B, Hawes R, Varadarajulu S. Non-superiority of lumen-apposing metal stents over plastic stents for drainage of walled-off necrosis in a randomised trial. Gut. 2019 Jul;68(7):1200-1209. doi: 10.1136/gutjnl-2017-315335. Epub 2018 Jun 1. PMID 29858393
- [Background] Kovacevic B, Vilmann P, Karstensen JG. Endoscopic Ultrasonography-Guided Gastrojejunostomies With Lumen-Apposing Metal Stents. Clin Gastroenterol Hepatol. 2017 Mar;15(3):459-460. doi: 10.1016/j.cgh.2016.09.144. Epub 2016 Sep 28. No abstract available. PMID 27693524
- [Derived] Karstensen JG, Novovic S, Hansen EF, Jensen AB, Jorgensen HL, Lauritsen ML, Werge MP, Schmidt PN. EUS-guided drainage of large walled-off pancreatic necroses using plastic versus lumen-apposing metal stents: a single-centre randomised controlled trial. Gut. 2023 Jun;72(6):1167-1173. doi: 10.1136/gutjnl-2022-328225. Epub 2022 Nov 29. PMID 36446550